CLINICAL TRIAL: NCT04646265
Title: The Effect of Non-surgical Periodontal Treatment on the Biomechanical Properties of the Periodontal Tissues, a Prospective Comparative Clinical Trial.
Brief Title: Effect of Periodontal Treatment on the Biomechanical Properties of the Periodontium.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bonn (Other)
Responsible Party: Principal Investigator, Karin Jepsen, Associated Professor, University of Bonn
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Ethik Nr.030/12
Record Dates: First submitted 2020-11-14; First posted 2020-11-27 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Periodontal Diseases
Keywords: Biomechanics; non-surgical periodontal treatment
MeSH Terms: conditions — Periodontal Diseases | interventions — Periodontal Index

STUDY DESIGN:
Intervention Model Description: prospective single center comparative clinical trial to investigate the biomechanical properties of periodontal tissues
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- periodontal treatment (Experimental): non-surgical root debridement
  Interventions: Other: periodontal treatment

INTERVENTIONS:
Other: periodontal treatment — non-surgical root debridement

SUMMARY:
Investigation of the biomechanical properties of the periodontal tissues in patients with periodontal disease. Non-surgical periodontal therapy will be assessed between baseline and 30 post-op by general clinical measurements (KT, PPD, CAL, BOP) as well as by biomechanical analysis and compared.

DETAILED DESCRIPTION:
The study is designed as a prospective single center comparative clinical trial to investigate the biomechanical properties of the periodontal tissues in 30 patients with periodontal disease.

Success of non-surgical periodontal therapy between baseline and 30 post-op will be assessed by general clinical measurements (KT, PD, CAL, BOP) as well as by biomechanical analysis. Besides assessment for regular treatment effectiveness, safety parameter such as wound healing and adverse events will be assessed.

Additionally 10 periodontally healthy persons without local inflammation and bone loss shall be monitored and used a control group for reference to the test teeth.

ELIGIBILITY:
Inclusion Criteria:

* Moderate/advanced/severe periodontitis
* Intact anterior dentition upper yaw.
* Expected performance of adequate oral hygiene
* Subjects must have voluntarily signed the informed consent form before any study related procedures
* Males and females with at least 18 years of age
* Subjects must be committed to the study and the required follow-up visits
* Subject must be judged in good general health as assessed by the investigator at time of non-surgical therapy

Exclusion Criteria:

* Any contraindications for subgingival instrumentation
* Uncontrolled diabetes or other uncontrolled systemic diseases
* Disorders or treatments that compromise wound healing
* Medical conditions requiring chronic high dose steroid therapy
* Bone metabolic diseases
* Radiation or other immuno-oppressive therapy
* Chronic anti-inflammatory treatment (≥3 times per week) within 4 weeks prior to treatment
* Presence of oral lesions (such as ulceration, malignancy)
* Mucosal diseases (e.g., lichen planus, mouth ulcer)
* History of malignant disease in the oral cavity or previous radiotherapy to the head or neck
* Treatment with an investigational drug or device within the 30 day period immediately prior to therapy on study day 0
* Female subjects who are nursing, pregnant, or plan to become pregnant
* Antibiotic treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Probing depth (PPD) at test tooth | 3 months
  mean PPD (mm)
Bleeding on Probing (BoP) | 3 months
  mean BoP (%)
Clinical attachment level (CAL) | 3 months
  mean attachment level (mm)
Biomechanical analysis | 3 months
  Tooth displacement (mm)

SECONDARY OUTCOMES:
Biotype/keratinized tissue width (KT) | 3 months
  mean - keratinized tissue width (KT)
1.General Oral Health Assessments Indices (GOHAI) | 3 months
  Limit the kinds of food - Questionaire by visual analogue scale (VAS)
2.General Oral Health Assessments Indices (GOHAI) | 3 months
  Trouble biting or chewing - Questionaire by visual analogue scale (VAS)
3.General Oral Health Assessments Indices (GOHAI) | 3 months
  Problems to swallow comfortably - Questionaire by visual analogue scale (VAS)
4.General Oral Health Assessments Indices (GOHAI) | 3 months
  Problems to speak clearly - Questionaire by visual analogue scale (VAS)
5.General Oral Health Assessments Indices (GOHAI) | 3 months
  Discomfort when eating any kind of food - Questionaire by visual analogue scale (VAS)
6.General Oral Health Assessments Indices (GOHAI) | 3 months
  Limit contact with people - Questionaire by visual analogue scale (VAS)
7.General Oral Health Assessments Indices (GOHAI) | 3 months
  Pleased with look of teeth- Questionaire by visual analogue scale (VAS)
8.General Oral Health Assessments Indices (GOHAI) | 3 months
  Used medication to relieve pain- Questionaire by visual analogue scale (VAS)
9.General Oral Health Assessments Indices (GOHAI) | 3 months
  Worried about teeth, gums or dentures - Questionaire by visual analogue scale (VAS)
10.General Oral Health Assessments Indices (GOHAI) | 3 months
  Self-conscious of teeth, gums or dentures - Questionaire by visual analogue scale (VAS)
11.General Oral Health Assessments Indices (GOHAI) | 3 months
  Uncomfortable eating in front of others - Questionaire by visual analogue scale (VAS)
12.General Oral Health Assessments Indices (GOHAI) | 3 months
  Sensitive to hot, cold or sweet foods - Questionaire by visual analogue scale (VAS)

CONTACTS AND LOCATIONS:
Overall Officials: Søren Jepsen, PhD, Principal Investigator — University of Bonn
Locations (1):
- Poliklinik für Parodontologie, Zahnerhaltung und Präventive Zahnheilkunde, Bonn, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Drolshagen M, Keilig L, Hasan I, Reimann S, Deschner J, Brinkmann KT, Krause R, Favino M, Bourauel C. Development of a novel intraoral measurement device to determine the biomechanical characteristics of the human periodontal ligament. J Biomech. 2011 Jul 28;44(11):2136-43. doi: 10.1016/j.jbiomech.2011.05.025. Epub 2011 Jun 15. PMID 21679952
- [Result] Keilig L, Drolshagen M, Tran KL, Hasan I, Reimann S, Deschner J, Brinkmann KT, Krause R, Favino M, Bourauel C. In vivo measurements and numerical analysis of the biomechanical characteristics of the human periodontal ligament. Ann Anat. 2016 Jul;206:80-8. doi: 10.1016/j.aanat.2015.08.004. Epub 2015 Sep 12. PMID 26395824
- [Result] Keilig L, Goedecke J, Bourauel C, Daratsianos N, Dirk C, Jager A, Konermann A. Increased tooth mobility after fixed orthodontic appliance treatment can be selectively utilized for case refinement via positioner therapy - a pilot study. BMC Oral Health. 2020 Apr 16;20(1):114. doi: 10.1186/s12903-020-01097-4. PMID 32299416
- [Result] Hajishengallis G. Periodontitis: from microbial immune subversion to systemic inflammation. Nat Rev Immunol. 2015 Jan;15(1):30-44. doi: 10.1038/nri3785. PMID 25534621
- [Result] Yoshida N, Koga Y, Peng CL, Tanaka E, Kobayashi K. In vivo measurement of the elastic modulus of the human periodontal ligament. Med Eng Phys. 2001 Oct;23(8):567-72. doi: 10.1016/s1350-4533(01)00073-x. PMID 11719079
- [Result] Jepsen S, Deschner J, Braun A, Schwarz F, Eberhard J. Calculus removal and the prevention of its formation. Periodontol 2000. 2011 Feb;55(1):167-88. doi: 10.1111/j.1600-0757.2010.00382.x. No abstract available. PMID 21134234